CLINICAL TRIAL: NCT03146871
Title: A Pilot/Safety Study of sEphB4-HSA in Combination With a Hypomethylating Agent (HMA) for Patients With Relapsed or Refractory Myelodysplastic Syndrome (MDS) and AML Previously Treated With a Hypomethylating Agent
Brief Title: Recombinant EphB4-HSA Fusion Protein and Azacitidine or Decitabine for Relapsed or Refractory Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia, or Acute Myeloid Leukemia Patients Previously Treated With a Hypomethylating Agent
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-16-6; NCI-2017-00623 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-16-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-04-25; First posted 2017-05-10 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Previously Treated Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine; Decitabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sEphB4-HSA, azacitidine, decitabine) (Experimental): Patients receive recombinant EphB4-HSA fusion protein intravenously (IV) over 60 minutes on days 1 and 15. Patients also receive azacitidine IV or subcutaneously (SC) on days 1-7 or days 1-5 and 8-9, or decitabine IV on days 1-5. Administration of recombinant EphB4-HSA fusion protein occurs before or after the HMA (not concurrently). Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Recombinant EphB4-HSA Fusion Protein

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Recombinant EphB4-HSA Fusion Protein — Given IV
  Other Names: sEphB4-HSA

SUMMARY:
This trial studies the side effects of recombinant EphB4-HSA fusion protein when given together with azacitidine or decitabine in treating patients with myelodysplastic syndrome, chronic myelomonocytic leukemia, or acute myeloid leukemia that has come back or has not responded to previous treatment with a hypomethylating agent. Recombinant EphB4-HSA fusion protein may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Hypomethylating agents, such as azacitidine and decitabine, slow down genes that promote cell growth and can kill cells that are dividing rapidly. Giving recombinant EphB4-HSA fusion protein together with azacitidine or decitabine may work better in treating patients with myelodysplastic syndrome, chronic myelomonocytic leukemia, or acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the toxicities and assess the tolerability of recombinant EphB4-HSA fusion protein (sEphB4-HSA) in combination with an approved hypomethylating agent (HMA) among patients with myelodysplastic syndrome (MDS) who are refractory to or have lost their response to one or more HMAs and among patients with relapsed/refractory acute myeloid leukemia (AML) previously treated with a HMA.

SECONDARY OBJECTIVES:

I. To measure the expression of EphB4 among marrow and peripheral blood blasts in patients with MDS & AML at baseline and over the course of treatment.

II. To measure the expression of immune check-point activating ligands (such as PD-L1, PD-L2) on marrow and peripheral blood blasts in patients treated with HMA and sEphB4-HSA in combination.

III. To profile immune subsets (activated and exhausted T cells, natural killer [NK] cells, T regulatory cells, and myeloid derived suppressor cells) in the peripheral blood and marrow in patients treated with HMA and sEphB4-HSA in combination.

IV. To assess efficacy of sEphB4-HSA in combination with an HMA as manifest by International Working Group (IWG) response criteria, as well as time to development of acute myeloid leukemia (AML) in patients with MDS and time to progression.

OUTLINE:

Patients receive recombinant EphB4-HSA fusion protein intravenously (IV) over 60 minutes on days 1 and 15. Patients also receive azacitidine IV or subcutaneously (SC) on days 1-7 or days 1-5 and 8-9, or decitabine IV on days 1-5. Administration of recombinant EphB4-HSA fusion protein occurs before or after the HMA (not concurrently). Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with advanced MDS requiring treatment with HMA and either refractory to at least 4 cycles or progressing after previously documented response

  * Patient must be treated within 6 months of the last HMA treatment and must be willing to be treated with the same agent they last received on this study
  * Prior treatment with novel HMA analog of decitabine on clinical trial is allowed; in such cases, decitabine will be used as the standard of care agent
* MDS classified as intermediate 1-risk or high risk according to the international prognostic scoring system (IPSS) or revised-IPSS
* Chronic myelomonocytic leukemia (CMML)
* Acute myeloblastic leukemia (AML) that was previously treated with HMA and is unfit for intensive chemotherapy

  * Patient must be within 6 months of prior treatment with HMA and must be willing to be treated with the same agent on this study
* During the 8 weeks prior to inclusion in study, subjects must have a baseline bone marrow examination including all of the following:

  * Cytomorphology to confirm bone marrow blasts
  * Cytogenetics
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Subject is able to understand and willing to comply with protocol requirements and instructions
* Subject has signed and dated informed consent
* Total bilirubin (except for Gilbert's syndrome) =< 2.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine =< 2.5 x ULN
* Women of childbearing potential (WOCBP) and male patients with WOCBP as partners must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of the investigational agent; subject is practicing an acceptable method of contraception (documented in case report form [CRF]); WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal; post menopause is defined as:

  * Amenorrhea >= 12 consecutive months without another cause or
* For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
* Women who are using oral contraceptives, other hormonal contraceptives (vagina products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential
* WOCBP must have a negative serum test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of investigational product
* Patients with uncontrolled hypertension

Exclusion Criteria:

* Patients with AML whose white blood cell count exceeds 25,000
* Corrected QT (QTc) (Fridericia Correction Formula) > 480 on electrocardiogram (ECG)
* Patients whose electrolytes (sodium, potassium, calcium, magnesium) are abnormal or cannot be normalized with standard intervention on the day of treatment with study drug
* Patients who are actively receiving any other anticancer therapy
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to HMAs
* Patients with a diagnosis of acute promyelocytic leukemia
* Patients with short life expectancy (less than 3 months) due to comorbidity other than MDS
* Female subjects who are nursing or pregnant (positive serum or urine Beta-human chorionic gonadotropin [B-hCG] pregnancy test)
* Patients with current alcohol or drug abuse
* Patients who have received treatment with an investigational drug within 30 days preceding the first dose of study medication
* Patients with uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients infected with hepatitis B, C or human immunodeficiency virus (HIV), unless they are on stable and effective antiviral treatment
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization; inhaled or topical steroids and adrenal replacement steroid doses > 10mg daily prednisone equivalent, are permitted in the absence of uncontrolled autoimmune disease
* MEDICATION-RELATED EXCLUSION CRITERIA
* Patients with uncontrolled hypertension (HTN) (> 160/90) will not be admitted onto the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 | Up to 30 days of the last dose of protocol treatment
  Will be tabulated and reported according to grade, type, cycle, and attribution.
Overall response defined as the occurrence of complete response, marrow complete response, partial response, or hematological improvement assessed by the IWG Working Group Criteria for MDS and AML | Up to 56 days (2 courses of protocol treatment)
  Will be calculated based on all patients who began treatment; exact 95% confidence intervals will be constructed.
Time to death from any cause | From start of treatment to death from any cause, assessed for up to 3 years
  Will be displayed with Kaplan-Meier plots.
Time to disease progression | From the start of treatment to the first disease progression or recurrence, assessed for up to 3 years
  Will be displayed with Kaplan-Meier plots.
Tolerability defined as the ability to complete two courses of treatment without the occurrence of dose limiting toxicity and the ability to begin course 3 within 4 weeks and graded according to the NCI CTCAE v4.0 | Up to 4 weeks following completion of course 2
  Will be tabulated and reported according to grade, type, cycle, and attribution.

OTHER OUTCOMES:
Change in the percent of bone marrow and peripheral blood blasts expressing EphB4 assessed by flow cytometry | Baseline up to 3 years
T-cell subset profile assessed by flow cytometry | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Casey O'Connell, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States